CLINICAL TRIAL: NCT06500793
Title: A Single and Multiple Dose Study to Evaluate the Pharmacokinetics of Oxycodone and PF614 When PF614 Capsule is Co Administered With Nafamostat as a Combination IR Solution and ER Capsule Formulation in Healthy Subjects
Brief Title: Single and Multi-Dose Study, Pharmacokinetics of Oxycodone and PF614 Co-Administered With Nafamostat (PF614-MPAR-102)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ensysce Biosciences (Industry)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: QSC301193
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — nafamostat

STUDY DESIGN:
Intervention Model Description: Single center, open-label study. Part 1 will assess impact of nafamostat (IR solution / ER beads) on oxycodone plasma levels when administered with 100 mg PF-614. Nafamostat will be increased from 1-10 mg if required to inhibit conversion of PF614 to oxycodone in an overdose situation (greater than 3 dose units taken simultaneously). Part 1 is intended to identify a nafamostat IR/ER combination that does not impact oxycodone release if 2 PF614 dose units are taken simultaneously yet show that nafamostat with 3 to 5 dose units inhibits conversion of PF614 to oxycodone in an OD situation (5 x 100 mg PF614 dose level). Results from Part 1 will define the dose units for Part 2 and 3. Part 2 will assess the impact of food on the exposure of PF-614 and nafamostat coadministered and PF-614 and nafamostat administered alone. Part 3 will assess multiple dosing (BID for 4.5 days) of 25 mg and 100 mg PF614 alone and co-administered with the selected nafamostat dose in the fasted state.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PF614 capsule with naltrexone HCl (Experimental): PF614 is an oxycodone prodrug. Part 1 doses = 100, 300 and up to 500 mg. Subjects will receive single daily doses at 5-14 days apart.
  Naltrexone, 50 mg Oral (Day -1, Day 1 and Day 2). All subjects will receive naltrexone block
  Interventions: Drug: PF614 capsule
- PF614 capsule concomitantly with nafamostat and naltrexone HCl (Experimental): PF614 is an oxycodone prodrug. Part 1 doses = 100, 300 and up to 500 mg. Nafamostat Mesylate is a trypsin inhibitor that blocks PF614 activation. Nafamostat IR solution (0.75 - XX mg); Nafamostat ER beads in capsule formulation (0.25 - YY mg) Naltrexone, 50 mg Oral (Day -1, Day 1 and Day 2). All subjects will receive naltrexone block
  Interventions: Drug: PF614 capsule; Drug: Nafamostat Mesylate

INTERVENTIONS:
Drug: PF614 capsule — PF614 capsules (25-100 mg)
  Other Names: PRF06104; Oxycodone prodrug
Drug: Nafamostat Mesylate — Nafamostat IR/ER solution/beads (total 1-10 mg)
  Other Names: Futhan
  Arms: PF614 capsule concomitantly with nafamostat and naltrexone HCl

SUMMARY:
A single and multiple-dose dose study to assess the pharmacokinetics (PK) of oxycodone, when PF614 is administered alone and with nafamostat as an immediate-release (IR) solution and/or extended-release(ER) capsule prototypes.

DETAILED DESCRIPTION:
PF614-MPAR is a combination of an oxycodone prodrug (PF614) and a protease inhibitor (nafamostat) that is intended to provide overdose protection when more than a prescribed dose may be taken simultaneously. A previous study (QSC203698) has explored various nafamostat formulations and identified an optimal combination of immediate release (IR) nafamostat and an extended release (ER) bead that when co-administered with 25 mg PF614 does not impact oxycodone exposure. However, when administered in an overdose situation (8 x unit dose level, 200 mg PF614 and 8 mg nafamostat), the nafamostat was able to inhibit trypsin which prevented the conversion of PF614 to oxycodone and hence prevented increased exposure of oxycodone when compared to 200 mg PF614 in the absence of nafamostat. The nafamostat formulation for the PF614 25 mg dose unit was identified 1 mg total nafamostat comprised of 0.75 mg IR and 0.25 mg ER beads (80:20 coating ratio). Ultimately the study defined the PF614-MPAR 25 mg dose unit.

Part 1 of the current study aims to define the PF614-MPAR 100 mg dose unit that is intended for commercialization, by exploring the impact of nafamostat on release of oxycodone from PF614 in naltrexone blocked healthy volunteers. Exposure of both oxycodone and PF614 will be evaluated following administration of 100 mg PF614-MPAR (PF614 and nafamostat (1 mg) as single dose unit or when administered up to 5 dose units simultaneously). If the nafamostat dose needs adjusting with 100 mg PF614, then this will also be assessed with the 50 mg PF614 dose unit in optional Part 1b. Part 1 will also assess exposure of a new 100 mg PF614 capsule formulation. In Part 2, the food effect will be assessed at the highest PF614 and nafamostat dose. If Part 1 is able to identify an appropriate PF614-nafamostat ratio then optional Part 3 will proceed which will investigate multiple dosing (twice a day dosing [BID] for 4.5 days) of 25 mg, and 100 mg PF614-MPAR optimized doses units (PF614 administered with the selected nafamostat unit dose) or PF614 alone to naltrexone blocked healthy volunteers in the fasted state.

The current study proposes to dose up to 500 mg PF614 (equivalent to 200 mg oxycodone); the 50 mg daily doses of naltrexone are anticipated to be more than sufficient to block 200 mg of an oxycodone-equivalent exposure.

ELIGIBILITY:
Inclusion Criteria:

1. Must be able to understand a written informed consent, which must be obtained prior to initiation of study procedures.
2. Must be willing and able to comply with all study requirements.
3. Aged 18 to 55 years, inclusive, at time of signing informed consent.
4. Must agree to use an adequate method of contraception (as defined in Section 9.4).
5. Healthy males or non pregnant, non lactating healthy females.
6. Body mass index (BMI) of 18.0 to 32.0 kg/m2 as measured at screening or, if outside the range, considered not clinically significant by the investigator.
7. Minimum weight of 50 kg at screening.

Exclusion Criteria:

1. Serious adverse reaction or serious hypersensitivity to any drug or formulation excipients.
2. Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hay fever is allowed unless it is active.
3. Significant serious skin disease, including rash, food allergy, eczema, psoriasis, or urticaria.
4. History of clinically significant cardiovascular, renal, hepatic, chronic respiratory or GI disease (Part 1 and Part 3 only: except cholecystectomy), gastrointestinal surgery (e.g. gastric bypass, gastric banding, colectomy), or neurological or psychiatric disorder, as judged by the investigator.
5. Subjects with a history of seizures.
6. Subjects with history of GI bleeding (excluding hemorrhoids) or history of peptic or duodenal ulcer disease.
7. Subjects with a history of bleeding disorders or coagulopathy.
8. Subjects with any personal history of arrhythmias or family history of significant cardiac disease (i.e., sudden death in first degree relative; myocardial infarction prior to 50 years old).
9. Part 2 only: Subjects with a history of cholecystectomy or gall stones.
10. Have poor venous access that limits phlebotomy.
11. Clinically significant abnormal clinical chemistry, hematology, coagulation or urinalysis as judged by the investigator (laboratory parameters are listed in Appendix 1). Subjects with Gilbert's Syndrome are allowed.
12. Subjects with a positive fecal occult blood test at screening or baseline (Part 3 only).
13. Subjects with a platelet count <150,000/µL or international normalized ratio >1.1 at screening.
14. Subjects with hemoglobin <LLN at screening and/or first admission.
15. Subjects with a QT interval corrected using Fridericia's formula (QTcF) above 450 msec at screening and/or first admission.
16. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) antibody results.
17. Positive serum pregnancy test at screening or first admission. Those who are pregnant or lactating will be excluded.
18. Subjects who have received any IMP in a clinical research study within 5 half lives or within 30 days prior to first dose. However, in no event shall the time between last receipt of IMP and first dose be less than 30 days.
19. Subjects who have previously been administered IMP in this study.
20. Subjects who are taking, or have taken, any prescribed or over the counter drug or herbal remedies (other than up to 4 g per day acetaminophen, HRT or hormonal contraception) in the 14 days before study treatment administration (see Section 11.4). Exceptions may apply on a case by case basis, if considered not to interfere with the objectives of the study, as determined by the investigator.
21. Subjects with an anticipated need for requiring aspirin, non-steroidal anti-inflammatory drugs, or anticoagulants in the 14 days after administration of the IMP.
22. History of any drug or alcohol abuse in the past 2 years.
23. Regular alcohol consumption in males >21 units per week and females >14 units per week (1 unit = 12 oz 1 bottle/can of beer, 1 oz 40% spirit, or 5 oz glass of wine).
24. A confirmed positive alcohol urine test at screening or first admission.
25. Current smokers and those who have smoked within the last 12 months.
26. Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months.
27. A confirmed positive urine cotinine test at screening or first admission.
28. Positive drug screen test result at screening or first admission (drug of abuse tests are listed in Appendix 1).
29. Male subjects with pregnant or lactating partners.
30. Donation of blood within 2 months or donation of plasma within 7 days prior to first dose of study treatment.
31. Subjects who are, or are immediate family members of, a study site or sponsor employee.
32. Failure to satisfy the investigator of fitness to participate for any other reason.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11-24 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-03-27 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic Tmax [Time to Maximum Plasma Concentration] | Parts 1 & 2 (PF614 single dose): predose, 0.25, 0.5, 1, 2, 4, 6, 12, 24, 36, 48, 72 hours. Part 3 (PF614 BID doses): Day 1 (predose, 0.25, 0.5, 1, 2, 4, 6, 12 hours; Days 2-3 (predose); Day 5 (predose, 0.25, 0.5, 1, 2, 4, 6, 12, 24, 36, 48, 72 hours)
  Time to maximum observed concentrations of oxycodone following administration of PF614 alone and with nafamostat
Pharmacokinetic Cmax [Maximum Plasma Concentration] | Parts 1 & 2 (PF614 single dose): predose, 0.25, 0.5, 1, 2, 4, 6, 12, 24, 36, 48, 72 hours. Part 3 (PF614 BID doses): Day 1 (predose, 0.25, 0.5, 1, 2, 4, 6, 12 hours; Days 2-3 (predose); Day 5 (predose, 0.25, 0.5, 1, 2, 4, 6, 12, 24, 36, 48, 72 hours)
  Maximum (peak) observed concentration of oxycodone following administration of PF614 alone and with nafamostat
Pharmacokinetic C24 [Plasma concentration at 24 hours] | Parts 1 & 2 (PF614 single dose): predose, 0.25, 0.5, 1, 2, 4, 6, 12, 24, 36, 48, 72 hours. Part 3 (PF614 BID doses): Day 1 (predose, 0.25, 0.5, 1, 2, 4, 6, 12 hours; Days 2-3 (predose); Day 5 (predose, 0.25, 0.5, 1, 2, 4, 6, 12, 24, 36, 48, 72 hours)
  Concentration of oxycodone at 24 hours post-dose following administration of PF614 alone and with nafamostat
Pharmacokinetic AUC(0-last) [Area Under the Curve] | Parts 1 & 2 (PF614 single dose): predose, 0.25, 0.5, 1, 2, 4, 6, 12, 24, 36, 48, 72 hours. Part 3 (PF614 BID doses): Day 1 (predose, 0.25, 0.5, 1, 2, 4, 6, 12 hours; Days 2-3 (predose); Day 5 (predose, 0.25, 0.5, 1, 2, 4, 6, 12, 24, 36, 48, 72 hours)
  Area under the concentration-time curve from time 0 to the time of last measurable concentrations of oxycodone following administration of PF614 alone and with nafamostat
Pharmacokinetic AUC(0-inf) [Area Under the Curve] | Parts 1 & 2 (PF614 single dose): predose, 0.25, 0.5, 1, 2, 4, 6, 12, 24, 36, 48, 72 hours. Part 3 (PF614 BID doses): Day 1 (predose, 0.25, 0.5, 1, 2, 4, 6, 12 hours; Days 2-3 (predose); Day 5 (predose, 0.25, 0.5, 1, 2, 4, 6, 12, 24, 36, 48, 72 hours)
  Area under the concentration-time curve from time 0 extrapolated to time-infinity of oxycodone following administration of PF614 alone and with nafamostat
Pharmacokinetic T1/2 [Half-life] | Parts 1 & 2 (PF614 single dose): predose, 0.25, 0.5, 1, 2, 4, 6, 12, 24, 36, 48, 72 hours. Part 3 (PF614 BID doses): Day 1 (predose, 0.25, 0.5, 1, 2, 4, 6, 12 hours; Days 2-3 (predose); Day 5 (predose, 0.25, 0.5, 1, 2, 4, 6, 12, 24, 36, 48, 72 hours)
  Terminal elimination half-life concentrations of oxycodone following administration of PF614 alone and with nafamostat

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Effects [Safety and Tolerability] | 30 Days
  Adverse events (AEs) including Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESIs), safety laboratory evaluations (hematology, coagulation, clinical chemistry, urinalysis), 12-lead electrocardiograms (ECGs), vital sign measurements, pulse oximetry and physical examinations.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Levy, MD, PhD, Principal Investigator — Medical Director, Quotient Sciences
Locations (1):
- Quotient Sciences, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kirkpatrick DL, Evans C, Pestano LA, Millard J, Johnston M, Mick E, Schmidt WK. Clinical evaluation of PF614, a novel TAAP prodrug of oxycodone, versus OxyContin in a multi-ascending dose study with a bioequivalence arm in healthy volunteers. Clin Transl Sci. 2024 Mar;17(3):e13765. doi: 10.1111/cts.13765. PMID 38511523
- [Background] Kirkpatrick DL, Schmidt WK, Morales R, Cremin J, Seroogy J, Husfeld C, Jenkins T. In vitro and in vivo assessment of the abuse potential of PF614, a novel BIO-MD prodrug of oxycodone. J Opioid Manag. 2017 Jan/Feb;13(1):39-49. doi: 10.5055/jom.2017.0366. PMID 28345745